CLINICAL TRIAL: NCT06714045
Title: Mediastinal Recurrence of Lympho-proliferative Disorders: a Biopsy is Needed
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MRLPD
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We would like to emphasise the need to perform a biopsy in patients with suspected persistence/recurrence of disease; the need to carefully plan the access route to minimise the risk of false negatives; the possibility of performing biopsies through all minimally invasive access routes available to the thoracic surgeon ensuring rapid clinical recovery and timely resumption of medical treatment in the event of recurrence.

DETAILED DESCRIPTION:
18 FDG PET is currently the gold standard for the staging of lymphoproliferative disorders such as lymphoma and a routine investigation for re-evaluation after first-line treatment; it is also a well-established re-evaluation modality in case of suspected disease recurrence.

Although FDG-PET/CT has an average sensitivity of 90% and a specificity of 91%, its diagnostic performance in combination with surgical biopsy has not yet been extensively evaluated.(1,2) The high predictive value of a negative PET scan, in the appropriate clinical context, helps to identify those patients with a complete metabolic response and therefore in complete remission.

In contrast, the persistence of metabolic activity (PET positivity) after systemic treatment cannot categorically confirm (or exclude) the presence (or absence) of viable lymphomatous tissue, due to the potential association of inflammatory reactions, which are normally manifested by increased hypercapture on PET scan.

For this reason, the persistence or reappearance of mediastinal hypermetabolic activity, in asymptomatic patients with no signs or symptoms of relapse, requires biopsy confirmation before making a diagnosis of disease relapse.

Current guidelines do not recommend the use of PET for the follow-up of patients in remission after lymphoma therapy due to its limited positive predictive value and considering the unequivocal correlation between hypermetabolic findings and definite disease relapse. However, an aggressive disease, in a district such as the mediastinum - where the rapid growth of a neoplastic disease may exacerbate symptoms of particular relevance due to the occupation of space or due to the infiltration of vital structures - may require a more thorough radiological follow-up including precisely the use of PET. Obviously, the discovery of a hypermetabolic finding in a completely asymptomatic patient requires histological confirmation of the relapse before making the definitive diagnosis of neoplastic recurrence.

For this reason, in these patients, the use of PET during follow-up helps to identify early metabolically suspicious lesions growing after remission from an aggressive neoplasm and to avoid, with timely therapeutic treatment, the appearance of particularly severe and sometimes extremely risky symptoms for the patient.

The finding of hypermetabolic mediastinal lesions, if the oncohaematologist recommends biopsy sampling, directs the surgeon to the most appropriate site for sampling considering that:

After treatment for lymphoma, coarse mediastinal masses with an inhomogeneous content (viable tissue alternating with necrotic tissue) and diffusely fibrotic often remain In the case of possible persistence of disease after first-line treatment, a voluminous mediastinal mass may be found on CT scan, while the hypermetabolic tissue (the site of suspected active lymphomatous residue) may be limited in size and sometimes focal.

Some lymphomatous diseases, at the time of relapse, may not be immediately identifiable by conventional radiology, particularly on CT scan, but may only be revealed by a functional investigation such as PET scan.

From a strictly surgical point of view, once the need to perform a biopsy has been established, the purely diagnostic nature of the procedure forces one to look for the least invasive access route, which is at low risk of complications and ensures a rapid convalescence.

The case history generated by a more than 20-year collaboration between the Seràgnoli Institute of the University Hospital and the Thoracic Surgery of the Maggiore Hospital in Bologna will be reviewed. The first 30 cases were published in 2007(3). Considering the lack of data in the reference literature, we will present the results of the review of the surgical approaches used in about 180 patients, the largest available case series on the subject.

ELIGIBILITY:
Inclusion Criteria:

Radiographic/scintigraphic suspicion of lymphoma persistence/recurrence after cytotoxic treatment Patients undergoing mediastinal biopsy procedure Obtaining informed consent.

Exclusion Criteria:

incomplete or missing data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent needle biopsy or surgical biopsy for suspected persistence or recurrence of lymphoma after cytotoxic treatment at the IRCCS Azienda Ospedaliero-Universitaria di Bologna Thoracic Surgery between 1 January 2002 and 31 January 2023
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2001-09-12 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
primary outcomes | 30 days after the surgery
  Verify the need for histological confirmation in patients undergoing cytotoxic therapy for lymphoma presenting radiological/scintigraphic signs of suspected persistence or mediastinal recurrence of disease.

SECONDARY OUTCOMES:
secondary outcomes | 30 days after the surgery
  Evaluate the sensitivity and specificity of the surgical techniques used to perform mediastinal biopsy sampling and assess the incidence of complications and hospitalisation times of each type of surgery: needle biopsy, mediastinoscopy, anterior mediastinotomy, cervico-manubriotomy, VATS and other more unusual surgical accesses, normally used in clinical practice for other pathologies as well, chosen from time to time on the basis of scintigraphic and radiological imaging in suspected lymphoma recurrence/persistence.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Nicola Forti Parri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna, Italy